CLINICAL TRIAL: NCT04494698
Title: Addressing Pain and Disability From Low Back Pain With an External Multimodal Neuromodulation Device
Brief Title: Impact of DuoTherm Compared to TENS on Pain and Disability With Acute and Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MMJ Labs LLC (Industry)
Collaborators: Sport and Spine Rehab Clinical Research Foundation (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Amy Lynn Baxter, Principal Investigator, MMJ Labs LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DuoTherm for Low Back Pain; 4R44DA049631 (NIH)
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Acute Low-back Pain; Chronic Low-back Pain; Pain, Intractable
Keywords: chronic low back pain; spine pain; medical device; analgesia; vibration; Multifidus
MeSH Terms: conditions — Pain, Intractable; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized active control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be instructed that non-drug interventions are being evaluated for their impact on opioid use and pain with low back pain, and that they will be self-assessing pain and reporting use of prescribed and over-the-counter medications. Study staff will train them on the device or TENS units via a pre-made video, but investigators and outcomes assessors (statistician) will not be informed of the hypothesis-driving condition arm. An assessment for blinding will be administered at the end of the data collection for participants, asking whether participants believe they are in treatment or control, and how confident they are.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DuoTherm VibraCool Back Device (Experimental): A multimodal low back pain relief device incorporating 8 mechanical stimulation patterns of vibration and 5 intensity settings with optional heat, cold, or pressure delivered through a sculpted metal plate attached by a belt and controlled by buttons on the belt. Patients will be instructed to use the device daily for 30 minutes.
  Interventions: Device: Duotherm VibraCool Back Device
- Multimodal TENS Unit (Active Comparator): LG SMART TENS stimulator is an 8-channel portable electrotherapy device featuring transcutaneous electrical nerve stimulation (TENS) therapeutic device, which is used for pain relief. The stimulator sends a gentle electrical current to underlying nerves and muscle groups via electrodes applied on the skin. The parameters of the device are controlled by buttons on a controller with an adjustable intensity level.
  Interventions: Device: TENS 8-channel unit

INTERVENTIONS:
Device: Duotherm VibraCool Back Device — Active New multimodal pain device
  Other Names: Vibracool plus heat or pressure; Buzzy
  Arms: DuoTherm VibraCool Back Device
Device: TENS 8-channel unit — LG Smart TENS unit
  Arms: Multimodal TENS Unit

SUMMARY:
Evaluate pain and disability change in Low Back Pain with DuoTherm Compared to Active Control

DETAILED DESCRIPTION:
160 patients with moderate to severe acute or exacerbations of chronic low back pain presenting for chiropractic and rehabilitation care will be randomized to one of two conditions: a pain relief belt device incorporating multiple speeds of vibration and optional heat, cold, and pressure delivered through a sculpted metal plate; or an 8 channel prescription TENS unit. Patients will be prompted by a Qualtrics text link to a secure data recording site collecting pain and medication use.

ELIGIBILITY:
Inclusion Criteria (same cohort as enrolled with NCT04491175):

* Presentation for treatment of acute or acute exacerbation of chronic low back pain
* Self-report NRS measures >=4 (moderate to severe)
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Willingness to communicate information on prescription pill # and dose, or dose and pill type if medication is prescribed by someone else.

Exclusion Criteria:

* Pacemaker
* Radicular pain likely reflecting a surgical or mechanical problem
* BMI greater than 50 (device won't fit, initially thought to be BMI 30 but up to 50 included)
* Sensitivity to cold or vibration (e.g Raynaud's or Sickle Cell Disease)
* Diabetic neuropathy rendering a patient unable to determine if the device is too hot
* New neurologic deficits
* Skin lesions over the low back area
* Contraindication to any medication for pain management that would impact analgesic use record
* Inability to apply DuoTherm or Active Control TENS Device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Change in current pain intensity from initial to final | Daily for 30 days, then weekly and monthly until 3 months (acute) or 6 months (chronic)
  Self-rated current pain on Numeric Rating Scale with 0 no pain and 10 maximum pain
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference | Baseline then weekly and monthly until 3 months (acute) or 6 months (chronic)
  Response formats for all scales are a 5-point ordinal rating scale of "Not at all," "A little bit," "Somewhat," "Quite a bit," and "Very much," where lower scores are better and higher scores indicate worse pain. The outcomes being addressed are Change in Monthly Pain Interference (8 questions, yielding possible scores of 8 (low) to 40 (highest) normed on a T-Score where 50 is the average in the United States, 40.7 is "no disability", 55 is mild, 57.7 is moderate, and 65.7 is severe

SECONDARY OUTCOMES:
Resolution of disability using PROMIS Pain Interference | Baseline then weekly and monthly until 3 months (acute) or 6 months (chronic)
  Achievement of average pain interference of a T-Score of 50 at last recorded PROMIS Pain Interference
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (8a) measures in those with intractable pain as defined and compared with surgical multifidus intervention studies | Initial through 6 month measurements (or 13 week if chronic enrolled as acute)
  Comparison between the experimental and active control interventions crosswalked with the Oswestry Disability outcomes in multifudus electrical stimulation studies.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Baxter, MD, Principal Investigator — Pain Care Labs (a dba of MMJ Labs)
Locations (2):
- United States (2):
  - Sport and Spine Rehab Clinics, Landover, Maryland
  - Sport and Spine Rehab Clinic, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the clinical results reported in any publications, after deidentification, will be available for a period of 36 months after publication to achieve approved aims of any researcher who provides a methodologically sound proposal. Proposals should be directed to info@mmjlabs.com. To gain acccess, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: up to 36 months after publication of results
Access Criteria: researchers providing approved methodologically sound proposals or requests

REFERENCES:
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, Delitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. Phys Ther. 2015 Feb;95(2):e1-e18. doi: 10.2522/ptj.2015.95.2.e1. PMID 25639530
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Stumbo SP, Yarborough BJ, McCarty D, Weisner C, Green CA. Patient-reported pathways to opioid use disorders and pain-related barriers to treatment engagement. J Subst Abuse Treat. 2017 Feb;73:47-54. doi: 10.1016/j.jsat.2016.11.003. Epub 2016 Nov 15. PMID 28017184
- [Background] Darnall BD, Colloca L. Optimizing Placebo and Minimizing Nocebo to Reduce Pain, Catastrophizing, and Opioid Use: A Review of the Science and an Evidence-Informed Clinical Toolkit. Int Rev Neurobiol. 2018;139:129-157. doi: 10.1016/bs.irn.2018.07.022. Epub 2018 Aug 6. PMID 30146045
- [Background] Furlan AD, Giraldo M, Baskwill A, Irvin E, Imamura M. Massage for low-back pain. Cochrane Database Syst Rev. 2015 Sep 1;2015(9):CD001929. doi: 10.1002/14651858.CD001929.pub3. PMID 26329399
- [Background] Maddalozzo GF, Kuo B, Maddalozzo WA, Maddalozzo CD, Galver JW. Comparison of 2 Multimodal Interventions With and Without Whole Body Vibration Therapy Plus Traction on Pain and Disability in Patients With Nonspecific Chronic Low Back Pain. J Chiropr Med. 2016 Dec;15(4):243-251. doi: 10.1016/j.jcm.2016.07.001. Epub 2016 Aug 25. PMID 27857632
- [Background] Cohen SP, Bhaskar A, Bhatia A, Buvanendran A, Deer T, Garg S, Hooten WM, Hurley RW, Kennedy DJ, McLean BC, Moon JY, Narouze S, Pangarkar S, Provenzano DA, Rauck R, Sitzman BT, Smuck M, van Zundert J, Vorenkamp K, Wallace MS, Zhao Z. Consensus practice guidelines on interventions for lumbar facet joint pain from a multispecialty, international working group. Reg Anesth Pain Med. 2020 Jun;45(6):424-467. doi: 10.1136/rapm-2019-101243. Epub 2020 Apr 3. PMID 32245841
- [Background] Tang X, Schalet BD, Hung M, Brodke DS, Saltzman CL, Cella D. Linking Oswestry Disability Index to the PROMIS pain interference CAT with equipercentile methods. Spine J. 2021 Jul;21(7):1185-1192. doi: 10.1016/j.spinee.2021.02.012. Epub 2021 Feb 19. PMID 33610807
- [Background] Gilligan C, Volschenk W, Russo M, Green M, Gilmore C, Mehta V, Deckers K, De Smedt K, Latif U, Sayed D, Georgius P, Gentile J, Mitchell B, Langhorst M, Huygen F, Baranidharan G, Patel V, Mironer E, Ross E, Carayannopoulos A, Hayek S, Gulve A, Van Buyten JP, Tohmeh A, Fischgrund J, Lad S, Ahadian F, Deer T, Klemme W, Rauck R, Rathmell J, Maislin G, Heemels JP, Eldabe S. Five-Year Longitudinal Follow-Up of Restorative Neurostimulation Shows Durability of Effectiveness in Patients With Refractory Chronic Low Back Pain Associated With Multifidus Muscle Dysfunction. Neuromodulation. 2024 Jul;27(5):930-943. doi: 10.1016/j.neurom.2024.01.006. Epub 2024 Mar 12. PMID 38483366
- [Background] Baxter AL, Thrasher A, Etnoyer-Slaski JL, Cohen LL. Multimodal mechanical stimulation reduces acute and chronic low back pain: Pilot data from a HEAL phase 1 study. Front Pain Res (Lausanne). 2023 Apr 26;4:1114633. doi: 10.3389/fpain.2023.1114633. eCollection 2023. PMID 37179530
- [Derived] Baxter AL, Etnoyer-Slaski JL, Tucker O, Williams JAR, Swartout K, Cohen LL, Lawson ML. Novel multimodal mechanical stimulation is superior to TENS to treat and prevent chronic low back pain: a randomized controlled trial. Front Pain Res (Lausanne). 2025 Aug 18;6:1625420. doi: 10.3389/fpain.2025.1625420. eCollection 2025. PMID 40901560

DOCUMENTS (1):
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT04494698/ICF_000.pdf